CLINICAL TRIAL: NCT01085539
Title: Oxygen Saturation Monitoring in the Neonatal Intensive Care Unit (NICU): An Observational Study of Response to Alarms
Brief Title: Oxygen Saturation Alarms in the Neonatal Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COV-M0-PO-A108
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Hypoxemia
Keywords: neonatal intensive care; infant pulse oximetry
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Infants will be observed in the neonatal intensive care unit for 4 hours. The observer will note the timing of oxygen saturation alarms, staff response, and interrupted staff activities.

DETAILED DESCRIPTION:
False alarms may be particularly prevalent in the neonatal intensive care unit (NICU) where uncontrolled motion of infants can intensify the problem. The performance of pulse oximeters is of particular importance in the NICU because of the danger that both hyperoxemia and hypoxemia pose to newborns; hyperoxemia can lead to chronic lung disease or retinopathy of prematurity, and hypoxemia depresses spontaneous ventilation. High false alarm rates contribute to the problem of noise in the NICU. They also have the potential to endanger patients if clinicians become inured to the continual alarms and ignore some that may be clinically relevant. There have been few studies on the utility of pulse oximeter alarms in the NICU, particularly with the new-generation technology. This study will build on the small body of existing literature on alarm rates in new-generation pulse oximeters in neonates and provide details about the relationship of the alarms to clinical interventions.

This is an observational study of 50 infants at three hospitals in the United States. The observer will be an experienced nurse with comprehensive training to ensure consistency. The infants and clinical staff will be observed for four hours continuously. Observers will note the timing of alarms, response, interrupted clinical staff activities, and any clinical interventions, and timing of interventions. Clinical staff will also be questioned on whether the alarm was consistent with a desaturation event. Infant characteristics may affect the frequency of alarms. Data collected will include age, gender, weight, ethnicity, diagnosis, and medications.

This study will evaluate the proportion of nuisance alarms relative to the proportion of clinically relevant alarms. It will also evaluate the differences in alarm frequencies across infant characteristics and characterize nurse activities interrupted by the alarms.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the NICU continuously monitored by pulse oximetry

Exclusion Criteria:

* Infants whose legal guardians do not consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: neonates in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Mecca, MD, Study Chair — Medtronic - MITG
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All infants in the neonatal intensive care unit that required continuous pulse oximetry qualified for the study during the dates of January 2010 through April 2010.
Groups:
- Infants With Oxygen Level Monitoring: In infants monitored for oxygen levels, the number of alarms that resulted in clinicians responding with an intervention that changed their care.
Period: Sat Secs Off--No Alarm Evaluation
Arm/Group | Infants With Oxygen Level Monitoring
Started | 50
Completed | 50
Not Completed | 0
Period: 10 Sat Secs--10 Second Alarm Evaluation
Arm/Group | Infants With Oxygen Level Monitoring
Started | 50
Completed | 50
Not Completed | 0
Period: 25 Sat Secs--25 Second Alarm Evaluation
Arm/Group | Infants With Oxygen Level Monitoring
Started | 50
Completed | 50
Not Completed | 0
Period: 50 Sat Secs--50 Second Alarm Evaluation
Arm/Group | Infants With Oxygen Level Monitoring
Started | 50
Completed | 50
Not Completed | 0
Period: 100Sat Secs-100 Second Alarm Evaluation
Arm/Group | Infants With Oxygen Level Monitoring
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infants With Oxygen Level Monitoring
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.73 (0.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Detection of Oxygen Alarms That Resulted in Clinicians Changing the Care of the Infant.
Description: Sat Secs is an oxygen alarm with 5 settings:0,10,25,50,and 100. At each setting,using the units of seconds,it filters nusiance alarms & identifies important alarms that result in the clinicians changing the care of the infant.
Time Frame: 4 hours
Population: All patients with complete data
Measure: Number; unit: percentage of interventions
Arm/Group | Infants With Oxygen Level Monitoring
Number analyzed (Participants) | 50
percentage of interventions
  Sat Secs Off | 39.9
  Sat Secs 10 | 44.4
  Sat Secs 25 | 48.0
  Sat Secs 50 | 50.3
  Sat Secs 100 | 53.2

ADVERSE EVENTS:
Arm/Group | Infants With Oxygen Level Monitoring
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
The study oximeter's detection could have been 60 seconds before or after the recorded clinical intervention because of sampling bias. There were many desaturations that led to alarms that had no interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less